CLINICAL TRIAL: NCT04368754
Title: Validity and Reliability the Turkish Version of the Oxford Participation and Activities Questionnaire (Ox-PAQ) in Older People
Brief Title: Validity and Reliability the Turkish Version of the Oxford Participation and Activities Questionnaire in Older People
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, MERV KARAPINAR, Research Assisstant, Physiotherapist, Hacettepe University
Other Study IDs: 191
Record Dates: First submitted 2020-04-26; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Healthy Aging
Keywords: Aged; Community Participation; Health; Physical Activity; Questionnaire
MeSH Terms: conditions — Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Patients evaluated with different questionnaire.

SUMMARY:
To evaluate the validity and reliability of Turkish version of the Oxford Participation and Activities Questionnaire (Ox-PAQ) for Turkish older population. Following the translation protocol of the Ox-PAQ, Short Form-12, Katz Index of Independence in Activities of Daily Living Scale, The Five Times Sit to Stand Test were administered to 230 older people. End of this study, occupational therapists, physiotherapists can use the it to assess activity and participation level of older people living in community

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Mini Mental State Examination score greater than 24,
* Able to mobilize independently.

Exclusion Criteria:

* Severe vision and hearing loss
* Having an orthopaedic, vestibular, neurological or mental problem
* Failure to cooperation
* Presence of an acute disease during recovery.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Older people (65 and older years)
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Ox-PAQ | One year
  It contains 23 items, each measured on a five-point Likert scale. Each of the 23 items is scored in the same direction (0=Never, 1=Rarely, 2=Sometimes, 3=Often, 4=Always). Also, Ox-PAQ consist of three domains, Routine Activities (14 items: nos. 1,2,3,4,5,6,7,8,9,10, 13,14,16,17), Social Engagement (4 items: nos. 11,12,15,18) and Emotional Well-Being (5 items: nos. 19,20,21,22,23). Raw scores of Ox-PAQ are transformed to a range from 0 to 100. The formula for scoring each dimension is as follows: sum of scores of each question in dimension/ ((4 x number of questions in dimension) x 100) (10). Higher scores reflect greater problems with activity and participation.

CONTACTS AND LOCATIONS:
Overall Officials: MERVE KARAPINAR, Principal Investigator — Suleyman Demirel University, Department of Physiotherapy and Rehabilitation
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karapinar M, Baskurt F, Baskurt Z, Gunal A, Kockar MC. Reliability and Validity of the Turkish Version of the Oxford Participation and Activities Questionnaire in Older People. Ann Geriatr Med Res. 2020 Dec;24(4):282-289. doi: 10.4235/agmr.20.0074. Epub 2020 Dec 24. PMID 33355854